CLINICAL TRIAL: NCT05514704
Title: Comparison of the Effects of Different Telerehabilitation Methods on Pain, Functional Limitation, Muscle Strength, Balance, and Quality of Life in Patients With Knee Osteoarthritis.
Brief Title: Effects of Different Telerehabilitation Methods on Pain, Functional Limitation, Muscle Strength, Balance, and Quality of Life in Patients With Knee Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eren Timurtas, PhD, Assoc Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2022.602/1
Record Dates: First submitted 2022-08-12; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation Group (Active Comparator): Synchronous Telerehabilitation Group will receive exercise therapy via video conference.
  Interventions: Other: Exercise Therapy via video conference
- Asynchronous Telerehabilitation Group (Experimental): Asynchronous Telerehabilitation Group will receive exercise therapy via mobile application.
  Interventions: Other: Exercise Therapy via mobile application

INTERVENTIONS:
Other: Exercise Therapy via video conference — The intervention will include the different levels of the following exercises that are given to the patient considering their functional level:
  1. Straight leg raise (Level 1-2-3)
  2. Quadriceps strengthening (Level 1-2-3)
  3. Hip abductor/adductor strengthening (Level 1-2-3)
  4. Hamstring stretch
  5. Gastrocnemius stretch
  Other Names: Therapeutic Exercise
  Arms: Synchronous Telerehabilitation Group
Other: Exercise Therapy via mobile application — The intervention will include the different levels of the following exercises that are given to the patient considering their functional level:
  1. Straight leg raise (Level 1-2-3)
  2. Quadriceps strengthening (Level 1-2-3)
  3. Hip abductor/adductor strengthening (Level 1-2-3)
  4. Hamstring stretch
  5. Gastrocnemius stretch
  Other Names: Therapeutic Exercise
  Arms: Asynchronous Telerehabilitation Group

SUMMARY:
The aim of our study is; To compare the effectiveness of asynchronous and synchronous telerehabilitation programs on pain, functional limitation, muscle strength, balance and quality of life parameters in patients with knee osteoarthritis.

60 patients with knee osteoarthritis who applied to Marmara University Faculty of Health Sciences Physiotherapy and Rehabilitation Department will be included in our study. The treatment and evaluations to be made will be explained and their consent will be obtained with their signatures. Patients will be randomly assigned to the asynchronous telerehabilitation group (n= 30 patients) and the synchronous telerehabilitation group (n= 30 patients). In the asynchronous telerehabilitation group, the rehabilitation program will be carried out via a mobile application (Diabetex). The coordinator will forward the exercise programs prepared specifically for the patients to the relevant participants through the application. On the other hand, telerehabilitation in the synchronous group will be carried out via video conference (Zoom). Patients will be taken to video conference calls and will perform their exercises simultaneously under the guidance of the researcher. An exercise program including lower extremity strengthening and stretching exercises will be applied to all patients. In both groups, the exercise program will be applied 3 days a week for 8 weeks, 1 session per day and 45 minutes per session. All outcome parameters will be evaluated by a blinded assessor who has not seen patients before. Patients starting the rehabilitation program will be evaluated at the beginning of the study, at weeks 4, 8, and 16.

The information of the patients participating in the study will be taken with the demographic data form. Pain in patients will be measured with the Visual Analog Scale, while the functionality of the patients will be evaluated with the WOMAC osteoarthritis index and the Lysholm Knee Scoring Scale. In addition, the affected quality of life of the patients will be evaluated with the Patient Generated Index and Short Form-12 scales. While the functional mobility of the patients was evaluated with the Timed Up and Go Test; functional capacities 2 Minute Walk Test, and lower extremity neuromuscular function levels 30 sec. It will be evaluated with Sit and Stand and 5 Sit and Stand performance tests. In addition, the Unilateral Posture Test, Limits of Stability Test, Sit and Stand Up Test will be performed using the NeuroCom Balance Master Posturography device for balance evaluation, and knee flexion and extension muscle strength and proprioception will be evaluated with the Isokinetic device.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative joint disease that occurs progressively in load-bearing joints under the influence of various mechanical, chemical and physical factors. Knee osteoarthritis, which is one of the most common musculoskeletal disorders in the world, causes functional limitation by causing symptoms such as edema, joint stiffness, crepitation, joint instability and deformity, especially pain. Traditional physiotherapy and rehabilitation approaches such as pharmacological agents, patient education, exercise, electrotherapy agents, and mobilization techniques are used in the conservative treatment of knee osteoarthritis. With the developing technology, telerehabilitation applications appear as an alternative approach to traditional physiotherapy. Telerehabilitation applications offer a convenient treatment option that is easily accessible, cost-effective, encourages the patient to repeat multiple and regular repetitions, and provides self-control by getting instant feedback. Telerehabilitation applications are divided into two; synchronous telerehabilitation, which allows exercising simultaneously with patients via video conference, and asynchronous telerehabilitation, where data and images are recorded via various mobile applications, and the patient can access exercise therapy when desired.

Although there are a limited number of studies investigating the effectiveness of telerehabilitation in patients with knee osteoarthritis in the literature, there is no study comparing asynchronous and synchronous telerehabilitation. Based on all this information, the aim of our study is; To compare the effectiveness of asynchronous and synchronous telerehabilitation programs on pain, functional limitation, muscle strength, balance and quality of life parameters in patients with knee osteoarthritis.

60 patients with knee osteoarthritis who applied to Marmara University Faculty of Health Sciences Physiotherapy and Rehabilitation Department will be included in our study. The treatment and evaluations to be made will be explained and their consent will be obtained with their signatures. Patients will be randomly assigned to the asynchronous telerehabilitation group (n= 30 patients) and the synchronous telerehabilitation group (n= 30 patients). In the asynchronous telerehabilitation group, the rehabilitation program will be carried out via a mobile application (Diabetex). The coordinator will forward the exercise programs prepared specifically for the patients to the relevant participants through the application. On the other hand, telerehabilitation in the synchronous group will be carried out via video conference (Zoom). Patients will be taken to video conference calls and will perform their exercises simultaneously under the guidance of the researcher. An exercise program including lower extremity strengthening and stretching exercises will be applied to all patients. In both groups, the exercise program will be applied 3 days a week for 8 weeks, 1 session per day and 45 minutes per session. All outcome parameters will be evaluated by a blinded assessor who has not seen patients before. Patients starting the rehabilitation program will be evaluated at the beginning of the study, at weeks 4, 8, and 16.

The information of the patients participating in the study will be taken with the demographic data form. Pain in patients will be measured with the Visual Analog Scale, while the functionality of the patients will be evaluated with the WOMAC osteoarthritis index and the Lysholm Knee Scoring Scale. In addition, the affected quality of life of the patients will be evaluated with the Patient Generated Index and Short Form-12 scales. While the functional mobility of the patients was evaluated with the Timed Up and Go Test; functional capacities 2 Minute Walk Test, and lower extremity neuromuscular function levels 30 sec. It will be evaluated with Sit and Stand and 5 Sit and Stand performance tests. In addition, the Unilateral Posture Test, Limits of Stability Test, Sit and Stand Up Test will be performed using the NeuroCom Balance Master Posturography device for balance evaluation, and knee flexion and extension muscle strength and proprioception will be evaluated with the Isokinetic device.

We think that the comparison of asynchronous and synchronous telerehabilitation methods, which can be preferred in the rehabilitation of a health problem such as knee osteoarthritis, which significantly affects the quality of life of individuals, causing high cost expenditures and loss of workforce, will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Pain less than or equal to 7 according to VAS
* Individuals aged 18-65
* Patients with independent mobility

Exclusion Criteria:

* Patients who have undergone surgery in the last 1 year
* Patients who have undergone total knee replacement or total hip replacement surgery
* Patients with acute trauma in the last 1 year
* Patients with uncontrolled chronic disease
* Patients who have received physical therapy in the last 6 months
* Patients who have received hyaluronic acid and corticosteroid injections in the last 6 months
* Patients with a respiratory condition that interferes with walking will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) osteoarthritis index | The WOMAC will be measured at baseline 2 minutes after pain assessment.
  The WOMAC osteoarthritis index is a 24-item scale that examines three dimensions: pain, stiffness, and physical function.
  Each question is scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated on its own and the total score ranges from 0 to 100. High scores indicate increased pain and stiffness and impaired physical function.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) osteoarthritis index | The WOMAC will be measured at the end of intervention (8. week) 2 minutes after pain assessment.
  The WOMAC osteoarthritis index is a 24-item scale that examines three dimensions: pain, stiffness, and physical function.
  Each question is scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated on its own and the total score ranges from 0 to 100. High scores indicate increased pain and stiffness and impaired physical function.
Visual analogue scale (VAS) | The pain will be measured at study entry (baseline) after inclusion.
  Pain will be measured using a 10 cm visual analogue scale (VAS). The participants places a mark on the line that best represented their perception of pain at that instant. The VAS score will be measured in cm from the left hand end of the line to the mark.
Visual analogue scale (VAS) | The pain will be measured at the end of intervention (8. week).
  Pain will be measured using a 10 cm visual analogue scale (VAS). The participants places a mark on the line that best represented their perception of pain at that instant. The VAS score will be measured in cm from the left hand end of the line to the mark.

SECONDARY OUTCOMES:
12-Item Short Form Survey (SF-12) | The SF-12 will be measured at baseline 2 minutes after WOMAC assessment.
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
  The SF-12 uses the same eight domains as the SF-36:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
12-Item Short Form Survey (SF-12) | The SF-12 will be measured at the end of intervention (8. week) 2 minutes after WOMAC assessment.
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. The SF-12 was created to reduce the burden of response.
  The SF-12 uses the same eight domains as the SF-36:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
30 Seconds Sit To Stand Test | The 30 Seconds Sit To Stand Test will be measured baseline 2 minutes after SF-12 assessment.
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults. The 30-Second Chair Test is administered using a folding chair without arms, with seat height of 17 inches (43.2 cm). The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving.
  The participant is seated in the middle of the chair, back straight; feet approximately a shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
  Have the patient practice a repetition or two before completing the test. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.
30 Seconds Sit To Stand Test | The 30 Seconds Sit To Stand Test will be measured at the end of intervention (8. week) 2 minutes after SF-12 assessment.
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults. The 30-Second Chair Test is administered using a folding chair without arms, with seat height of 17 inches (43.2 cm). The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving.
  The participant is seated in the middle of the chair, back straight; feet approximately a shoulder width apart and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest.
  Have the patient practice a repetition or two before completing the test. If a patient must use their arms to complete the test they are scored 0. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.
2 Minute Walk Test | The 2 Minute Walk Test will be measured at baseline 5 minutes after 30 Seconds Sit To Stand Test assessment.
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity.
  The person is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured.
  Start timing when the individual is instructed to "Go". Stop timing at 2 minutes. Assistive devices can be used but should be kept consistent and documented from test to test.
  If physical assistance is required to walk, the test should not be performed. The measuring wheel is helpful to determine the distance walked. The person should walk at the fastest speed possible. Rest breaks are allowed if needed.
  Before starting the test, the observer gives initial instructions :
2 Minute Walk Test | The 2 Minute Walk Test will be measured at the end of intervention (8. week) 5 minutes after 30 Seconds Sit To Stand Test assessment.
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity.
  The person is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured.
  Start timing when the individual is instructed to "Go". Stop timing at 2 minutes. Assistive devices can be used but should be kept consistent and documented from test to test.
  If physical assistance is required to walk, the test should not be performed. The measuring wheel is helpful to determine the distance walked. The person should walk at the fastest speed possible. Rest breaks are allowed if needed.
  Before starting the test, the observer gives initial instructions :
Quadriceps and Hamstring Muscle Strength | The Quadriceps and Hamstring Muscle Strength will be measured at baseline 15 minutes after 2 Minute Walk Test assessment.
  Isometric muscle strength of the Quadriceps Femoris and Hamstring muscle groups will be measured at 30º and 60º using the Biodex® System Pro3 (Biodex Corp. Shirley NY, USA) isokinetic test dynamometer. During the test, the back angle of the dynamometer seat is adjusted to 85° and the patients are asked to hold on to the bars next to the seat. The leg to be tested is fixed with the help of belts to prevent compensation of the pelvis and trunk. The test protocol was explained to the patients beforehand; They were instructed to apply force (30º and 60º angle) to the specified area of the device with as much effort as they could and not to allow the device to move their extremities. Before the isometric muscle strength test is performed on the isokinetic system, the patients were given 3 repetitive exercises. The dynamometric test was first performed with 3 repetitions at an angle of 30º, and then 3 repetitions at 60º. 15 seconds between tests, rest periods are given.
Quadriceps and Hamstring Muscle Strength | The Quadriceps and Hamstring Muscle Strength will be measured at the end of intervention (8. week) 15 minutes after 2 Minute Walk Test assessment.
  Isometric muscle strength of the Quadriceps Femoris and Hamstring muscle groups will be measured at 30º and 60º using the Biodex® System Pro3 (Biodex Corp. Shirley NY, USA) isokinetic test dynamometer. During the test, the back angle of the dynamometer seat is adjusted to 85° and the patients are asked to hold on to the bars next to the seat. The leg to be tested is fixed with the help of belts to prevent compensation of the pelvis and trunk. The test protocol was explained to the patients beforehand; They were instructed to apply force (30º and 60º angle) to the specified area of the device with as much effort as they could and not to allow the device to move their extremities. Before the isometric muscle strength test is performed on the isokinetic system, the patients were given 3 repetitive exercises. The dynamometric test was first performed with 3 repetitions at an angle of 30º, and then 3 repetitions at 60º. 15 seconds between tests, rest periods are given.

IPD SHARING:
Plan to Share IPD: No